CLINICAL TRIAL: NCT03676543
Title: Mutual Interactions Between Absence Epilepsy Seizures and the Integration of Sensory Stimuli
Acronym: Absence SLI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This is the end of the inclusion period and only 1 patient has been recruited.
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCX_2017_28
Record Dates: First submitted 2018-07-31; First posted 2018-09-18 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Childhood or Juvenile Absence Epilepsy
MeSH Terms: conditions — Epilepsy, Absence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Timed repetitive sensory stimulation (Experimental): Timed repetitive sensory stimulation (TRSS) will be applied at the onset or during seizures
  Interventions: Procedure: Timed repetitive sensory stimulation

INTERVENTIONS:
Procedure: Timed repetitive sensory stimulation — Timed repetitive sensory stimulation (TRSS) will be applied at the onset or during seizures

SUMMARY:
Epileptic seizures arise from neuronal defects that often alter the capacity of the brain to process sensory information. During absence seizures, a frequent epileptic syndrome in children, the normal conscious and perceptual processes are temporarily interrupted. This is the result of abnormal synchronized neural activities in the thalamo-cortical loops, leading to bilateral spike-and-wave discharges (SWDs) in the cortical electroencephalograms (EEGs). The brain mechanisms underlying the lack of sensory experience during absence seizures are disputed. Based on preliminary data, the investigators hypothesize that the alternation of 'spike' and 'wave' patterns during seizure could cause a time-to-time inconstancy in cortical responsiveness, preventing conscious perception. Using a real-time closed-loop stimulation system, the investigators will research how the S- and W-patterns specifically alter the sensory-evoked responses in the EEG. During a standard EEG, visual stimulations will be applied between and during absence seizures to test the hypothesis that repeated sensory stimuli, applied with an appropriate timing relative to the seizure-related oscillatory cycle, could negatively interfere with the regenerative network mechanisms involved in the occurrence of SWDs. The completion of this project should permit to unveil a new neuronal mechanism supporting the lack of conscious experience during absences and pave the way for new clinical non-invasive strategies to interrupt ongoing seizure activity.

ELIGIBILITY:
Inclusion criteria :

* Age 2-20 years
* childhood or juvenile absence epilepsy defined by International Ligue Against Epilepsy (ILAE)
* Electroencephalogram (EEG) indicated for clinical follow-up

Non inclusion criteria:

* Visual deficit
* Abnormal Magnetic Resonance Imaging (MRI)
* Medical history of photosensitive epileptic seizures

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Modification of the frequency within the peak-wave complexes according to the repeated sensory stimulation and the duration of the absence epilespy crisis | 1 hour
  Modification of the frequency within the peak-wave complexes according to the repeated sensory stimulation and the duration of the absence epilespy crisis
Modification of the duration of the absence epilespy crisis according to the repeated sensory stimulation | 1 hour
  Modification of the duration of the absence epilespy crisis according to the repeated sensory stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation OPH A. de Rothschild, Paris, France